CLINICAL TRIAL: NCT03072290
Title: Comparison of Different Dose of Steroid Injection in Carpal Tunnel Syndrome
Brief Title: Corticosteroid Injection in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-07-006A
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Triamcinolone Acetonide; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose steroid (Experimental): ultrasound-guided steroid injection using 1ml of 10 mg (10mg/ml) triamcinolone acetonide (Shincort) mixed with 1 ml of 2% lidocaine hydrochloride (Xylocaine)
  Interventions: Drug: Triamcinolone Acetonide; Drug: lidocaine hydrochloride
- comparator (Active Comparator): ultrasound-guided steroid injection using 1ml of 40 mg (40mg/ml) triamcinolone acetonide (Shincort) mixed with 1 ml of 2% lidocaine hydrochloride (Xylocaine)
  Interventions: Drug: Triamcinolone Acetonide; Drug: lidocaine hydrochloride

INTERVENTIONS:
Drug: Triamcinolone Acetonide — ultrasound-guided injection using 1ml of 10 mg (10mg/ml) or 40 mg (40 mg/ml) triamcinolone acetonide (Shincort)
  Other Names: triamcinolone acetonide 10mg/ml (shincort, YSP, Taiwan)
Drug: lidocaine hydrochloride — ultrasound-guided injection using 1 ml of 2% lidocaine hydrochloride (Xylocaine)
  Other Names: lidocaine hydrochloride (Xylocaine)

SUMMARY:
To compare the effectiveness of different dose of ultrasound guided steroid injection in patient with carpal tunnel syndrome, by using clinical and electrophysiological parameters in evlauation

DETAILED DESCRIPTION:
This is a prospective, single-blinded randomized controlled study to determine the efficacy of low dose corticosteroid in patient with CTS. Patient with CTS were randomly assigned to group receiving ultrasound guided steroid injection with different dosage of triamcinolone acetonide (Shincort) mixed, 1ml 10mg (10mg/ml) or 1ml 40mg (40mg/ml) with 1 ml of 2% lidocaine hydrochloride. The follow up at 6 and 12 weeks includes Boston Carpal Tunnel Questionnaire, nerve conductive study and VAS pain score.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CTS
* The diagnosis of CTS was confirmed by electrophysiological tests.

Exclusion Criteria:

* presence of thenar atrophy
* existence of disorders such as hypothyroidism, diabetes mellitus, chronic renal failure, or rheumatoid arthritis; any accompanying orthopedic or neurologic disorders that could mimic CTS such as cervical radiculopathy, polyneuropathy, proximal median nerve entrapment, or thoracic outlet syndrome
* prior steroid injection into the affected carpal tunnel within 6 months or ever received carpal tunnel surgery
* history of distal radius fracture
* pregnancy or lactation
* regular use of systemic NSAIDs ,corticosteroids or diuretics
* known allergy to corticosteroids and local anesthetics.
* impaired cognitive function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-18 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the scores on the Boston Carpal Tunnel Questionnaire (BQ). | at 6, 12 weeks
  The BQ was interviewed-administered to assess the severity of symptoms and functional status.

SECONDARY OUTCOMES:
Change from Baseline in Median nerve distal motor latency | at 6, 12 weeks
  the CMAPs were obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode was placed on the muscle belly, and the reference electrode was placed on the tendon insertion. The median nerve was stimulated 8 cm proximal to the active recording electrode. Distal motor latencies were measured from the onset of stimulus artifact to the onset of the CMAP
Change from Baseline in sensory nerve conduction velocity | at 6, 12 weeks
  SNAPs were obtained using an antidromic method and recorded by surface electrodes placed at the proximal and distal interphalangeal joints of the index finger for the median nerve and the same joints of the little finger for the ulnar nerve. The median nerves were stimulated at the wrist at a distance of 14 cm from the wrist to the active electrode. Distal sensory latencies were measured from the onset of the stimulus artifact to the onset of the SNAP. SNCV was calculated dividing the distance of 14 cm by the distal sensory latency.
Change from Baseline in compound muscle action potential amplitude (CMAP) | at 6, 12 weeks
  the CMAPs were obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode was placed on the muscle belly, and the reference electrode was placed on the tendon insertion. The median nerve was stimulated 8 cm proximal to the active recording electrode. The amplitude of CMAP were measured from baseline to negative peak.
Change from Baseline in self-reported pain intensity | at 6, 12 weeks
  Patients were asked to indicate the intensity of their average level of pain for the wrist-hand region within the past 1 week, using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei veteran general hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu PC, Liao KK, Lin KP, Chiu JW, Wu PY, Chou CL, Wang NY, Wang JC. Comparison of Corticosteroid Injection Dosages in Mild to Moderate Idiopathic Carpal Tunnel Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Nov;101(11):1857-1864. doi: 10.1016/j.apmr.2020.06.018. Epub 2020 Jul 16. PMID 32682938